CLINICAL TRIAL: NCT05686707
Title: Characterization of Different Phenotypes of Microvascular Dysfunction and Their Impact on Angina Severity in Patients With Chronic Angina in the Absence of Obstructive Coronary Artery Disease
Acronym: MiVa
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Collaborators: University of Catanzaro (Other); I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other); Università degli Studi di Ferrara (Other); IRCCS Multimedica (Other); Università di Siena (Unknown); University of Parma (Other); Universita di Verona (Other); Ospedale Policlinico San Martino (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); A.O.U. Città della Salute e della Scienza (Other); Azienda Policlinico Umberto I (Other); Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Giovanni Esposito, Full Professor, Federico II University
Other Study IDs: 333-21
Record Dates: First submitted 2022-07-18; First posted 2023-01-17 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Angina CCS Classe II-IV - IMR, RFR, FFR,CFR
Keywords: CCS IMR, RFR, FFR,CFR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study will be to identify different phenotypes of microvascular dysfunction and their associations with the severity of anginal symptoms assessed through the Seattle Angina Questionnaire(SAQ-7).

DETAILED DESCRIPTION:
After administration of unfractionated heparin (100UI/Kg), a special pressure guide (Pressure Wire X, Abbott), equipped with a distal sensor capable of measuring pressure and temperature, will be introduced inside the anterior descending branch (IVA) of the left coronary artery and hyperemia will be induced by intravenous infusion of adenosine. The IMR will be calculated using the thermodilution technique, and is given by the product between the mean distal pressure, in the left anterior descending coronary artery, and the mean transit time (Tmn) during maximal hyperemia.

During the procedure, additional coronary physiological indices will be calculated such as:

* Quiescent full cycle flow ratio (RFR), - Fractional flow reserve (FFR),
* Coronary flow reserve (CFR)

In order to identify different phenotypes of microvascular dysfunction, as follows:

* Phenotype A: Patients with IMR>25, CFR <2 and FFR>0.80 (concordant pure-microvascular pathological results)
* Phenotype B: patients with IMR>25, CFR>2 and FFR>0.80 (increased microvascular hyperemic resistance, maintenance of microvascular reactivity)
* Phenotype C: Patients with IMR 25, CFR 2 and FFR>0.80 (normal hyperemic resistance and reduced reactivity) All these phenotypes can also be combined with pathological FFR measures (<0.80) (phenotypes A1, B1, C1).

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria will be considered for study participation:

Age ≥18 and <85 years. Chronic coronary syndrome (including patients with anginal equivalents) Angina CCS class II-IV Evidence of inducible reversible ischemia in noninvasive trials

Availability of the following measurements:

* Microvascular resistance index (IMR)
* Quiescent full cycle flow ratio (RFR),
* fractional flow reserve (FFR),
* Coronary flow reserve (CFR) Willingness to participate and sign the informed consent document prior to the procedure.

Exclusion Criteria:

At least one of the following:

Pregnancy or breastfeeding. Medical or psychological conditions that would compromise proper and orderly participation.

Left ejection fraction less than 30% Prior coronary artery bypass surgery (CABG) Decompensated congestive heart failure (CHF) Chronic or acute renal failure with creatinine >2mg/dl Severe valve disease Patients with comorbidities limiting life expectancy to less than one year.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes, aged between 18 and 85 years, with clinical indication to perform a diagnostic coronary angiography, according to the current guidelines of the European Society of Cardiology will be enrolled. (ESC)
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
(SAQ-7) | 12 months
  Identify different phenotypes of microvascular dysfunction and their associations with anginal symptom severity assessed through the Seattle Angina Questionnaire (SAQ-7).

SECONDARY OUTCOMES:
characterization of the severity of angina | 12 months
  To validate the ability of the microvascular resistance index to identify patients who have microvascular disease and its utility in characterizing angina severity. Identify different phenotypes of microvascular dysfunction and their associations with comorbidities, cardiovascular risk factors, and drug therapy. A sub-analysis on the use of different antianginal drugs will be performed to better understand the impact of pharmacotherapy on different microvascular dysfunction phenotypes.
  Evaluate the health status of patients in different microvascular dysfunction phenotypes through the EQ-5D-5L questionnaire.
  EQ-5D is a standardized measure of health status developed by the EuroQoL Group in order to provide a simple and generic measure of health for clinical and economic evaluation.
  Evaluate the state of depression induced by the disease through "The Brief Illness Perception Questionnaire (B-IPQ).

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University of Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: No